CLINICAL TRIAL: NCT04500938
Title: Cardiac Mitochondrial Function in Explanted Human Hearts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Roni Nielsen, Principal Investigator, University of Aarhus
Other Study IDs: 0404-92-02062020
Record Dates: First submitted 2020-07-22; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: End-stage Heart Failure
Keywords: Mitochondrial function; High Resolution Respirometry; Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endomyocardial biopsies taken from the explanted heart after removal during heart transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Treatment of heart failure has improved considerably in the past decades. Despite this improvement, the disease may progress into an end-stage ultimately leaving the physicians with no other treatment option than heart transplantation (HTx). There are multiple etiologies underlying heart failure. Cardiomyopathy is the leading cause for HTx in any age-group with coronary artery disease being the second most common cause in adult patients.

Alterations in the mitochondrial function have been recognized as key factors in heart failure.

During the transplant procedure the diseased heart is removed, providing a unique opportunity to collect samples eligible for thorough mitochondrial examination.

Hopefully, the knowledge gained from this investigation will contribute with important insights in the diseased myocardial energy metabolism. Such knowledge may pave the way for development of treatments targeting both energy substrate supply for adenosine-triphosphate generation produced by the mitochondria as well as mitochondrial function in the failing heart.

Hypothesis:

The pathological myocardial function seen in heart failure is related to dysfunctional cardiac mitochondria

Objective:

To examine if cardiac mitochondrial function in end-stage heart failure of multiple etiologies is inferior to mitochondrial function in transplanted hearts with no signs of rejection or vasculopathy.

Design:

Myocardial mitochondrial function analyzed from 24 explanted hearts will be compared to endomyocardial biopsies from 20 HTx patients at scheduled biopsies (1 or 2 years after implantation).

DETAILED DESCRIPTION:
Background:

Treatment of heart failure has improved considerably in the past decades. Despite this improvement, the disease may progress into an end-stage ultimately leaving the physicians with no other treatment option than heart transplantation (HTx). There are multiple etiologies underlying heart failure. Cardiomyopathy is the leading cause for HTx in any age-group with coronary artery disease being the second most common cause in adult patients.

Alterations in the mitochondrial function have been recognized as key factors in heart failure. The understanding of the complex interaction of the mitochondria in regulation of the metabolism and cellular apoptosis has brought new perspectives to research in heart failure. It is now known that the myocardial mitochondrial density changes and their function and integrity is impaired during heart failure.

During the transplant procedure the diseased heart is removed, providing a unique opportunity to collect samples eligible for thorough mitochondrial examination.

The collected myocardial tissue samples will be evaluated with High Resolution Respirometry, examining the glucose coupled respiratory capacity of permeabilized myocardial fibers. The respiratory capacity in the diseased fibers will be compared to the respiratory capacity in fibers from coronary healthy HTx patients transplanted 1 to 2 years prior to acquisition of the fibers.

Hopefully, the knowledge gained from this investigation will contribute with important insights in the diseased myocardial energy metabolism. Such knowledge may pave the way for development of treatments targeting energy substrate supply for adenosine-triphosphate generation produced by the mitochondria as well as mitochondrial function in the failing heart.

Hypothesis:

The pathological myocardial function seen in heart failure is related to dysfunctional cardiac mitochondria.

Objective:

To examine if cardiac mitochondrial function in end-stage heart failure of multiple etiologies is inferior to mitochondrial function in transplanted hearts with no signs of rejection or vasculopathy.

Design and Endpoint:

Myocardial mitochondrial function analyzed from 24 explanted hearts will be compared to endomyocardial biopsies from 20 HTx patients at scheduled biopsies (1 or 2 years after implantation).

Endpoints: 1) Mitochondrial respiratory capacity. 2) Mitochondrial complex function, outer membrane integrity and mitochondrial content.

Methods:

High-resolution respirometry:

High-resolution respirometry is used to measure mitochondrial respiratory capacity in endomyocardial biopsies. After appropriate preparation, two biopsies are transferred to an oxygraph (Oxygraph-2k; Oroboros, Innsbruck, Austria) for high resolution respirometry. Mitochondrial respiratory capacity will be analyzed in a step-by-step manner using titrations of substrates and inhibitors to evaluate glucose coupled respiration in the fibers. High-resolution respirometry analysis is performed within 8 hours after the biopsy has been taken.

After analysis the tissue will be snap-frozen in liquid nitrogen and stored in a research biobank at -80 degrees celsius until examination of citrate synthase activity is carried out. Hereafter, any remaining tissue will be destroyed.

Electron microscopy:

A sample from each biopsy used for high-resolution respirometry will be used for electron microscopy (EM) to evaluate mitochondrial volume density (MitoVD) and integrity. Muscle samples are fixated for 24 hours in glutaraldehyde and washed 4x15 minutes with Na-cacodylate buffer before being casted in Epon. The Epon casted tissue will be stored in a research biobank until EM analysis. Ultra-thin sections of the Epon-blocks (60 nm) are cut in three depths and dyed with uranyl acetate and lead citrate. Imaging is performed with an EM 208 transmission electron microscope and a Megaview III camera. All fibers are photographed at 10.000 × magnification in a randomized order. MitoVD is estimated from mitochondrial fractional area and only distinct fibers will be used in the final analysis.

Statistics:

Normally distributed data will be presented as mean ± standard deviation; non-normally distributed data will be presented as median and interquartile range. Categorical data are presented as absolute values or percentages. Histograms and Q-Q plots will be used to check continuous values for normality. Between-group differences will be assessed by t-test for normally distributed data and Mann-Whitney U test for non-normally distributed data. Statistical significance at a p-value of <0.05.

Sample size calculation:

At present there are no test-retest evaluation of mitochondrial respiratory analysis in endomyocardial biopsies from explanted human hearts. However, a recent study performed at our department on myocardial biopsies demonstrated that a total sample size of 40 human subjects in a 1:1 parallel group design was able to identify differences between the two groups (unpublished data).

Data collection and processing:

Source data will be recorded in the patient's electronic patient record or on specific worksheets.

A centralized electronic Case Report Form (CRF) will be constructed for data capture. Data will be stored until completion of the project, after which, it will be transmitted to the Danish Data Archives.

Perspectives:

HTx is the golden standard treatment for patients suffering from end-stage heart failure, but its limitations cannot be ignored. Firstly, the procedure is accompanied by a substantial risk and a significant percentage of patients suffer from acute graft failure. Furthermore, HTx patients have a higher risk of severe infections and cancer, and up to 50% of HTx patients suffer from cardiac allograft vasculopathy 10 years after transplantation, all of which are highly related to mortality. Hence, postponing HTx is desirable, if health and life-quality can be kept at an acceptable level. In this context, mitochondrial function seems to be pivotal, as approaches to assess mitochondrial function in the failing heart may prove to pave the way for new follow-up algorithms and even treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from the recipient

Exclusion Criteria:

* Myocardial biopsy from the explanted heart not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All heart transplanted patients, transplanted at Aarhus University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-08-30 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
State 2 respiration (GM) | Within 5 minutes.
  Complex I-linked respiration, induced by Malate and Glutamate.
State 3 respiration (GM3) | Within 10 minutes.
  Complex I-linked respiration with adenosine diphosphate (ADP), induced by Malate, Glutamate and ADP.
State 3 respiration (GMS3) | Within 15 minutes.
  Complex I+II-linked respiration, induced by Malate, Glutamate, ADP and Succinate.
State 4 respiration (4o) | Within 30 minutes.
  Complex I+II-linked respiration not linked to adenosine triphosphate production, induced by inhibition of complex V by Oligomycin.
Residual Oxygen Consumption (ROX) | Within 45 minutes.
  Respiration not linked to the electron transport chain, induced by inhibition of complex I by Rotenone, complex III by Antimycin A and complex V by Oligomycin.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Eiskjær, MD, DMSc, Principal Investigator — University of Aarhus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb S, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Heart Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1244-54. doi: 10.1016/j.healun.2015.08.003. Epub 2015 Aug 28. No abstract available. PMID 26454738
- [Background] Murphy E, Ardehali H, Balaban RS, DiLisa F, Dorn GW 2nd, Kitsis RN, Otsu K, Ping P, Rizzuto R, Sack MN, Wallace D, Youle RJ; American Heart Association Council on Basic Cardiovascular Sciences, Council on Clinical Cardiology, and Council on Functional Genomics and Translational Biology. Mitochondrial Function, Biology, and Role in Disease: A Scientific Statement From the American Heart Association. Circ Res. 2016 Jun 10;118(12):1960-91. doi: 10.1161/RES.0000000000000104. Epub 2016 Apr 28. PMID 27126807
- [Background] Jespersen NR, Yokota T, Stottrup NB, Bergdahl A, Paelestik KB, Povlsen JA, Dela F, Botker HE. Pre-ischaemic mitochondrial substrate constraint by inhibition of malate-aspartate shuttle preserves mitochondrial function after ischaemia-reperfusion. J Physiol. 2017 Jun 15;595(12):3765-3780. doi: 10.1113/JP273408. Epub 2017 Feb 27. PMID 28093764
- [Background] Gormsen LC, Svart M, Thomsen HH, Sondergaard E, Vendelbo MH, Christensen N, Tolbod LP, Harms HJ, Nielsen R, Wiggers H, Jessen N, Hansen J, Botker HE, Moller N. Ketone Body Infusion With 3-Hydroxybutyrate Reduces Myocardial Glucose Uptake and Increases Blood Flow in Humans: A Positron Emission Tomography Study. J Am Heart Assoc. 2017 Feb 27;6(3):e005066. doi: 10.1161/JAHA.116.005066. PMID 28242634
- [Background] Brown DA, Perry JB, Allen ME, Sabbah HN, Stauffer BL, Shaikh SR, Cleland JG, Colucci WS, Butler J, Voors AA, Anker SD, Pitt B, Pieske B, Filippatos G, Greene SJ, Gheorghiade M. Expert consensus document: Mitochondrial function as a therapeutic target in heart failure. Nat Rev Cardiol. 2017 Apr;14(4):238-250. doi: 10.1038/nrcardio.2016.203. Epub 2016 Dec 22. PMID 28004807
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Dipchand AI, Benden C, Christie JD, Dobbels F, Kirk R, Rahmel AO, Yusen RD, Stehlik J; International Society for Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: Thirtieth Official Adult Heart Transplant Report--2013; focus theme: age. J Heart Lung Transplant. 2013 Oct;32(10):951-64. doi: 10.1016/j.healun.2013.08.006. No abstract available. PMID 24054804